CLINICAL TRIAL: NCT04937751
Title: Multicenter Study on Invasive Fusariosis : Looking for Markers of Infection and Resistance
Brief Title: Markers of Infection and Resistance in Invasive Fusariosis
Acronym: FUSIMIR
Status: Recruiting | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Anne DEBOURGOGNE, Principal investigator, Central Hospital, Nancy, France
Other Study IDs: 2020PI202
Record Dates: First submitted 2021-06-16; First posted 2021-06-24 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Fusariosis
MeSH Terms: conditions — Fusariosis | interventions — Environmental Biomarkers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and fungal strains
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Invasive fusariosis
  Interventions: Diagnostic Test: biomarkers
- Fusarium keratitis
  Interventions: Diagnostic Test: biomarkers

INTERVENTIONS:
Diagnostic Test: biomarkers — galactomannan, betaDglucan, resistance markers

SUMMARY:
In recent decades, invasive fusarioses have been emerging fungal pathologies with high mortality. The prognosis depends on the speed of the diagnosis, but currently biological diagnosis is mainly based on fungal culture, no specific biomarker for this microorganism is available in current clinical practice. The genus Fusarium also shows reduced sensitivity to antifungals commonly used and recommended in clinical practice, such as voriconazole or amphotericin B.

The main objective of this study is to describe the proportions of different fungal species in positive fungal cultures in patients with invasive fungal infection (IFI) or fungal keratitis. The secondary objectives are the description of the dosage of galactomannans, beta (1,3) -D-glucans and the rate of detection of DNA circulating in case / control groups for the 2 clinical forms studied. In patients with evidence of Fusarium wilt, the study will describe the distribution of the different minimum inhibitory concentrations (MIC) depending on whether or not different antifungals are taken, the vital status at 3 months, and the response or not to treatment. Finally, the presence of genetic markers will be described according to the groups of MIC values.

ELIGIBILITY:
Inclusion Criteria:

* Suspicion of invasive fungal infection involving the performance of a blood culture or a skin biopsy or diagnosis of keratitis involving the taking of a cornea sample
* Fungal culture carried out on this sample
* Person having been informed of the research and not having opposed the use of their data

Exclusion Criteria:

* Clinical diagnosis of superficial fusarium wilt (onychomycosis, etc.)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will have 2 parts:
  1. a first descriptive section carried out through a study of 2 cohorts of patients (patients suspected of IFI / with a diagnosis of keratitis) for whom a fungal culture is carried out;
  2. a second descriptive part (then potentially comparative if the statistical power is sufficient) carried out through 2 case-control studies nested in each of the patient cohorts (patients suspected of IFI / with a diagnosis of keratitis): these studies will consist of a population of cases (patients with Fusarium wilt) and 1 or 2 populations of controls (patients with negative culture on the one hand and patients with positive culture for a fungus of another genus in Fusarium on the other hand for invasive fusarioses).
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-07-19 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
proportions of different fungal species in positive fungal cultures in patients with invasive fungal infection (IFI) or fungal keratitis | 2021-2026

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU Nancy, Vandœuvre-lès-Nancy, France